CLINICAL TRIAL: NCT02897856
Title: Efficacy and Safety of Intramuscular Midazolam Compared to Buccal Midazolam in Pediatric Seizures: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Intramuscular Midazolam Compared to Buccal Midazolam in Pediatric Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, DR. KHALID AL-ANSARI, Senior consultanat, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-00050
Record Dates: First submitted 2016-09-04; First posted 2016-09-13 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buccal midazolam (Active Comparator): Study subject will receive buccal midazolam and intramuscular placebo. The dose of buccal midazolam is 0.3 mg/kg
  Interventions: Drug: Buccal midazolam
- intramuscular midazolam (Active Comparator): Study subject will receive intramuscular midazolam and buccal placebo. The dose of intramuscular midazolam is 0.25 mg/kg.
  Interventions: Drug: Intramuscular midazolam

INTERVENTIONS:
Drug: Buccal midazolam — Study subject will receive Buccal midazolam, Intramuscular placebo.
  Arms: Buccal midazolam
Drug: Intramuscular midazolam — Study subject will receive Intramuscular midazolam,Buccal placebo
  Arms: intramuscular midazolam

SUMMARY:
The goal of this study is to prove that intramuscular midazolam is more effective than buccal midazolam in cessation of seizure activity with comparable side effects.

DETAILED DESCRIPTION:
Both buccal and intramuscular midazolam have been used to control seizures with variable succuss rates and side effects.

In this study the investigators are going to assign patient randomly to receive either buccal or intramuscular midazolam. Then will compare both efficacy and side effect in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 month to 14 years who will be presented to the pediatric emergency or attended by emergency medical service who have active seizure and had no intravenous access would be eligible for the study.

Exclusion Criteria:

* Cardiac arrest
* Head trauma
* Drowning
* Congenital heart disease
* Inborn errors of metabolism
* Electrolyte imbalance (hypocalcaemia, hyponatremia and hypoglycemia)
* Hemodynamic instability
* Allergy to benzodiazepines
* Focal seizures with preserved level of consciousness

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Cessation of seizure activity five minutes after treatment with study medication. | five minutes
  Cessation of abnormal motor activity with regaining of consciousness.

SECONDARY OUTCOMES:
Major side effects. | 2 hours after cessation of seizures.
Duration of seizure. | 5 minutes
Recurrence of seizure activity within one hour after treatment with study medication. | one hour

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No